CLINICAL TRIAL: NCT02801968
Title: Tap Block and Cesarean Delivery: Efficacy and Consumption of Postoperative Drugs
Acronym: TAPFANS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: S. Anna Hospital (Other)
Responsible Party: Principal Investigator, Ilaria Farinelli, Doctor, S. Anna Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIIAV1574
Record Dates: First submitted 2016-05-28; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Cesarean Delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tap block (Experimental): Tap block with ropivacaine 2 mg/kg at the end of cesarean delivery. Postoperative analgesia with acetaminophen and tramadol plus NSAIDs (nonsteroidal anti-inflammatory drugs) as rescue dose.
  Interventions: Procedure: Tap block; Other: intravenous analgesia
- control group (Active Comparator): Postoperative analgesia after cesarean delivery with acetaminophen and tramadol plus NSAIDs (nonsteroidal anti-inflammatory drugs) as rescue dose.
  Interventions: Other: intravenous analgesia

INTERVENTIONS:
Procedure: Tap block
  Arms: Tap block
Other: intravenous analgesia

SUMMARY:
The purpose of this study is to determine the efficacy of Tap block after cesarean delivery as a component of multimodal analgesia and evaluation of postoperative drugs consumption.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* written consent
* anesthesiologist's assent on preoperative evaluation

Exclusion Criteria:

* age< 18 years
* uncooperative patients
* written consent not obtained
* local anesthetic allergy
* BMI > 35

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Pain evaluation with Numerical Rating Scale (NRS) | Pain evaluation with NRS at 2,6,12,24 hours after cesarean delivery in TAP block group and in the control group.
  We don't want to measure the change between each assessment within a single group, instead we want considering the difference in the measurements between two separate groups (TAP block group and control group) for each time point.

SECONDARY OUTCOMES:
Evaluation of NSAIDs (nonsteroidal anti-inflammatory drugs) consumption as rescue dose during the first 24 hours after cesarean delivery | Doses of NSAIDs (nonsteroidal anti-inflammatory drugs) administered at 2, 6, 12 ,24 hours after cesarean delivery TAP block group and in the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Osepdale Santa Maria delle Croci, Ravenna, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No